CLINICAL TRIAL: NCT03701789
Title: Evaluation of Bone Quality in Patients With Rheumatoid Arthritis Treated With Baricitinib: Single Centre, Mode of Action Study (BARE BONE)
Brief Title: Effect of Baricitinib Treatment on Peripheral Bone in RA
Acronym: BAREBONE
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BAREBONE2018
Record Dates: First submitted 2018-10-04; First posted 2018-10-10 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Rheumatoid Arthritis; Bone Density; Finger Joints
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Rheumatoid Arthritis (Other): In-label treatment with Baricitinib
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Baricitinib — Effect of Baricitinib on vBMD measured by HR-pQCT
  Other Names: Oliumiant

SUMMARY:
Patients with Rheumatoid Arthritis (RA) suffer systemic and peripheral bone loss. In this study we aim to test the efficacy of in-label treatment with Baricitinib on the volumetric bone mineral density in patients with RA over 52 weeks. Inclusion of RA patients comprises pathologic volumetric bone mineral density measured by (High Resolution peripheral quantitative Computed Tomomgraphy) HR-pQCT maging of finger joints.

DETAILED DESCRIPTION:
Systemic and local bone loss is a pathognomonic feature of rheumatoid arthritis and can be seen in a very early phase of the disease. Understanding the pathogenesis of rheumatoid arthritis (RA) has advanced substantially in recent years. The mode of action of immunosuppressive medication on pro-inflammatory cytokines, different cell types or activation of cells is intensively studied and understood. In contrary, little is known on how these medications influence bone damage in peripheral joints in terms of bone density, bone microstructure, bone quality or erosions. This is due to different reasons. One factor is the lack of suitable, user-independent imaging tools for outcome measurements. For example, using conventional X-ray of the hand and fingers, no information can be obtained about the volumetric density, microarchitecture, bone quality or volumetric erosion size. Applying Dual-energy Xray absorptiometry (DXA) of peripheral joints, does also not provide information about the volumetric bone density and no accurate difference can be obtained regarding cortical or trabecular density parameters. Magnetic Resonance Imaging (MRI) as an outcome measure in RA enables good the detection and partly quantification of erosions, however no information about bone density can be quantified. HR-pQCT (high resolution peripheral quantitative computed tomography) imaging allows in detail (82 micrometer isotropic voxelsize) evaluation of density, microstructure parameters as well as quantification of erosions in peripheral joints. Furthermore, HR-pQCT data allows the biomechanical analysis of the bone and therefore statements on the bone quality can be made.

Modulating inhibitors targeting the Janus Kinase (JAK) - Signal Transducer and Activator of Transcription (STAT) pathway, effect pro-inflammatory cytokines and have been approved for therapy in RA patients. Analysis of the inhibition of the JAK-STAT pathway in rheumatoid arthritis synovium showed decreased phosphorylation of STAT1. Also pro-inflammatory activation of STAT1 and downstream targets were inhibited by JAK inhibition. More interesting, STAT1-/- mice have higher bone density due to Runx2 activation but are otherwise are indistinguishable from wildtype mice . Furthermore, inhibition of STAT1 accelerates bone repair after trauma, a similar process in our observation in rheumatoid arthritis joints. On the other hand, JAK1 deficient mice showed reduced body mass peri-natal which has been speculated to indicate bone growth delays. Focusing on bone loss, JAK inhibition (tofacitinib) suppressed osteoclast mediated bone destruction via reduction of T cell derived RANKL. In vitro we observed that osteoclast (OC) differentiation was not influenced by JAK inhibition in regard to OC numbers and transcription factor expression. Interestingly, in osteoblast cultures, JAK inhibition induced Runx2, Col1a and Osterix. In co-culture assays with osteoblasts and OC precursors JAK inhibition led to decreased OC differentiation.Thus JAK inhibition mediated OC function is not only influenced by T cell but also osteoblast derived RANKL and therefore interferes in the balance of bone turnover by activating osteoblasts.Using HR-pQCT measurements of fingers of RA patients treated with tofacitinib in a small sample size we detected an astonishing gain of volumetric bone mineral density (mg Hydroxylapatite/mm³). Furthermore, we noticed a decrease of the intra-articular cortical porosity and a positive change of erosion size. In these cases, volumetric bone density in metacarpal joints improved up to 20 %. In our experience, regarding other immunosuppressive medication for example anti-TNF Inhibition, no comparable effect was observed.

The longitudinal setup of this mode of action study is used to determine the effect of baricitinib on the change of the volumetric bone mineral density in RA patients with pathologic vBMD measured by HR-pQCT technique over 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Main inclusion criteria:

Patients eligible for inclusion in this study have to fulfil all of the following criteria:

* Subject must be able to understand and communicate with the investigator and comply with the requirements of the study, must give a written and signed and dated informed consent before any study assessment is performed
* Male or non-pregnant, non-lactating female subjects aged between 18 - 74
* Women of childbearing potential must oblige to use a highly effective method of birth control until at least 4 weeks after the last IMP administration
* Diagnosis of RA according to the ACR/EULAR criteria and with symptoms for at least 3 months with moderate to severe RA
* pathologic volumetric bone density, microstructure or presence of erosions detected by HR-pQCT and or MRI measurement
* Previous treatment with at least one DMARD (e.g. methotrexate) without sufficient clinical response or stopped due to toxicities
* Fulfil criteria for baricitinib treatment according to its SmPC

Exclusion Criteria:

* Ongoing pregnancy status or breast-feeding

  * Chest X-ray or chest MRI with evidence of ongoing infectious or malignant process, obtained within 3 months or according to local guidelines, prior to screening and evaluated by a qualified physician
  * Contraindication for baricitinib treatment according to its SmPC
  * Current treatment with bDMARDs or other JAK-inhibitors
  * Creatinine clearance < 60ml/min (calculated analogue MDRD)
  * Current treatment with OAT3 inhibitors
  * History or evidence of ongoing alcohol or drug abuse, within the last six months before inclusion
  * Participation in an interventional clinical trial with an IMP within the last 4 weeks

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2021-10-11 (Estimated); Study Completion 2021-10-11 (Estimated)

PRIMARY OUTCOMES:
Change in volumetric bone mineral density (vBMD) in metacarpal and radial bone between baseline and week 52 in patients with rheumatoid arthritis treated with baricitinib as determined by HR-pQCT | 52 weeks
  HR-pQCT

CONTACTS AND LOCATIONS:
Overall Officials: Arnd Kleyer, MD, Principal Investigator — Department of Internal Medicine 3, Rheumatology and Immunology Universital Hospital Erlangen
Locations (1):
- Universitiy Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Simon D, Minopoulou I, Kemenes S, Bayat S, Tascilar K, Mutlu MY, Valor-Mendez L, Kronke G, Hueber AJ, Schett G, Kleyer A. Baricitinib Improves Bone Properties and Biomechanics in Patients With Rheumatoid Arthritis: Results of the Prospective Interventional BARE BONE Trial. Arthritis Rheumatol. 2023 Nov;75(11):1923-1934. doi: 10.1002/art.42617. Epub 2023 Sep 21. PMID 37229650